CLINICAL TRIAL: NCT00165711
Title: The Role of Methycobalamin in Early Dementia Patients With Vitamin B12 Deficiency and Hyperhomocysteinaemia.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AS-006 (MBL-HKG-05-01); NCT00164983 (obsolete NCT alias)
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2019-02-19 (Actual); Status verified 2005-12

CONDITIONS: Dementia With Vitamin B12 Deficiency
MeSH Terms: interventions — mecobalamin

INTERVENTIONS:
Drug: Mecobalamin

SUMMARY:
Patients who fit the inclusion criteria are admitted into the study. They are given 3 IV injection of MBL in the first week and one tablet three times a day for 16 weeks.

ELIGIBILITY:
Inclusion:

* Patients with Dementia
* Serum B12 < 200 pmol/l
* Serum Homocysteine level > 11.0 micro mol/L

Exclusion:

Significant communication problems

* deafness, dysarthria, dysphasia etc.
* unstable DM or hypertension
* alcohol abuse
* co-existing diseases which may affect cognition e.g. cognitive cardiac failure, respiratory failure
* folate < 10 g/dl
* haemoglobin concentration < 10g/d
* abnormal thyroid function test or VDRL

Min Age: 60 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2003-03

PRIMARY OUTCOMES:
Mattis dementia rating scale

SECONDARY OUTCOMES:
Category fluency test
Delirium rating scale
CNPI
MMSE
Plasma homocysteine
Plasma isoprostane

CONTACTS AND LOCATIONS:
Overall Officials: Romeo Chu, Study Director — Eisai Asia Regional Services Ltd.
Locations (1):
- Chinese University of Hong Kong, Hong Kong, Hong Kong, China